CLINICAL TRIAL: NCT05991765
Title: Evaluation of Digit Tip and Split Skin Donor Site Transcriptome
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University Hospital Schleswig-Holstein (Other)
Responsible Party: Principal Investigator, Tobias Kisch, Principal Investigator, University Hospital Schleswig-Holstein
Other Study IDs: DigitTip2023
Record Dates: First submitted 2023-08-07; First posted 2023-08-15 (Actual); Last update posted 2023-08-15 (Actual); Status verified 2023-08

CONDITIONS: Digit Tip Wound; Split Skin Donor Site
Keywords: Digit Tip; Split Skin Donor Site; Transcriptome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Digit Tip Wound: Experimental Wound Exudate from Digit Tip Wounds
  Interventions: Other: Digit Tip Wound
- Split Skin Donor Site Wound: Active Comparator Wound Exudate from Split Skin Donor Site Wound
  Interventions: Other: Split Skin Donor Site Wound

INTERVENTIONS:
Other: Digit Tip Wound — Digit Tip Wound Exudate Sample Collected while Dressing Change
  Groups: Digit Tip Wound
Other: Split Skin Donor Site Wound — Split Skin Donor Site Wound Exudate Sample while Dressing Change
  Groups: Split Skin Donor Site Wound

SUMMARY:
Regrowth of amputated fingertips presents a unique regenerative healing process in mammals, with subcutaneous volume regrowth, restoration of the dactylogram, and suppression of scar formation. In addition, wound healing from split-thickness donor sites shows almost scar-free healing. Transcriptome analysis is necessary to better understand the specific healing mechanisms of these two wound entities. Since no data are available to date, this study aims to fill the gap.

DETAILED DESCRIPTION:
Regrowth of amputated fingertips presents a unique regenerative healing process in mammals, with subcutaneous volume regrowth, restoration of the dactylogram, and suppression of scar formation. In addition, wound healing from split-thickness donor sites shows almost scar-free healing. Transcriptome analysis is necessary to better understand the specific healing mechanisms of these two wound entities. Since no data are available to date, this study aims to fill the gap.

ELIGIBILITY:
Inclusion Criteria:

1. Digit Tip Wound: Wound Exudate from healthy patients: Consent-capable patients ≥18 years of age with clean Digit Tip Wound
2. Split Skin Donor Site Wound: Wound Exudate from healthy patients: Consent-capable patients ≥18 years of age with clean Split Skin Donor Site Wound

Exclusion Criteria:

* Inflammation
* Borderline
* Infectious Disease

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Consent-capable patients ≥18 years of age with either Digit Tip Wound or Split Skin Donor Site
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Differences in RNA-Expression pattern | 5 Weeks
  Differences in RNA-Expression pattern between Digit Tip Wound and Split Skin Donor Site Wound

CONTACTS AND LOCATIONS:
Locations (1):
- University of Schleswig-Holstein, Lübeck, Schleswig-Holstein, Germany